CLINICAL TRIAL: NCT00227461
Title: Levetiracetam (Keppra) to Improve Chronic Aphasia in Post-stroke Patients.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kessler Foundation (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Principal Investigator, A. M. Barrett, MD, Director, Stroke Rehabilitation Research, Kessler Foundation
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AMBarrett1; none applicable
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Aphasia; Stroke
Keywords: Aphasia; Stroke
MeSH Terms: conditions — Aphasia; Stroke | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wait control (Other): Levitiracetam is started after a delay, with dosage and administration as described below.
  Interventions: Drug: Levetiracetam first, then wait
- Treatment first (Experimental): Levitiracetam is started immediately after baseline data is collected; dosage and administration as described below.
  Interventions: Drug: Wait first, then levetiracetam

INTERVENTIONS:
Drug: Wait first, then levetiracetam — Levetiracetam 250 mg orally twice daily for 7 days. This will increase to 500 mg oral twice daily for 7 days the following week. If this dose is tolerated, it will then be increased to 750 mg orally twice daily for another 7 days and then increased to 1000 mg orally twice daily for 7 days.
  Other Names: Keppra
  Arms: Treatment first
Drug: Levetiracetam first, then wait — subjects with aphasia will take levetiracetam and we will evaluate their speech, language, and memory in an ABAB design
  Other Names: Keppra
  Arms: Wait control

SUMMARY:
The study investigates the possibility that levetiracetam may improve the symptoms of chronic post-stroke aphasia.

DETAILED DESCRIPTION:
In the study, 50 post-stroke subjects with aphasia will take levetiracetam and we will evaluate their speech, language, and memory in an ABAB design.

ELIGIBILITY:
Inclusion Criteria:

* Stroke
* Aphasia
* Can give consent

Exclusion Criteria:

* Renal failure
* Pregnancy
* Other neurological condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-09 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Speech and language assessment | 6 months - 1year

SECONDARY OUTCOMES:
Memory assessment | 6 months to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: A.M. Barrett, MD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States